CLINICAL TRIAL: NCT06829030
Title: Comparıson Of The Effectıveness Of Intramuscular Dıclofenac Sodıum And Subcutaneous 5% Dextrose Injectıon In Patıents Applyıng To The Emergency Department Wıth Low Back Paın.
Brief Title: Comparison of the Efficacy of Diclofenac Sodium and Subcutaneous 5% Dextrose Injection in Low Back Pain.
Acronym: NPT
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, huseyin mutlu, Ass.Prof., Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: AksarayUTRH-1
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain, Mechanical
Keywords: Low back pain; neuroprolotherapy; , diclofenac sodium,; emergency department
MeSH Terms: conditions — Low Back Pain; Emergencies | interventions — Diclofenac

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided into two groups. The first group will receive subcutaneous 5% dextroseprolotherapy, and the second group will receive intramuscular 75 mg diclofenac sodium injection.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- %5 dekstroz proloterapi (Experimental): The study is planned to include 75 volunteer patients with low back pain who presented to the emergency department of Aksaray University Education and Research Hospital. The first group will receive subcutaneous 5% dextrose prolotherapy (approximately 75 patients), and the second group will receive intramuscular 75 mg diclofenac sodium injection.
  Interventions: Drug: 5% dextrose prolotherapy
- intramuscular 75 mg diclofenac sodium injection (Active Comparator): The study is planned to include 75 volunteer patients with low back pain who presented to the emergency department of Aksaray University Education and Research Hospital. The first group will receive subcutaneous 5% dextrose prolotherapy (approximately 75 patients), and the second group will receive intramuscular 75 mg diclofenac sodium injection.
  Interventions: Drug: Diclofenac 75mg/ml

INTERVENTIONS:
Drug: 5% dextrose prolotherapy — The first group will receive subcutaneous 5% dextrose prolotherapy (approximately 75 patients), and the second group will receive intramuscular 75 mg diclofenac sodium injection
  Other Names: Diclofenac 75mg/ml
  Arms: %5 dekstroz proloterapi
Drug: Diclofenac 75mg/ml — The first group will receive subcutaneous 5% dextrose prolotherapy (approximately 75 patients), and the second group will receive intramuscular 75 mg diclofenac sodium injection (approximately 75 patients).
  Other Names: 5% dextrose prolotherapy
  Arms: intramuscular 75 mg diclofenac sodium injection

SUMMARY:
The aim was to compare the effectiveness of intramuscular diclofenac sodium and subcutaneous 5% dextrose injection in patients presenting to the emergency department with low back pain using the visual analog scale (VAS).

DETAILED DESCRIPTION:
The aim was to compare the effectiveness of intramuscular diclofenac sodium and subcutaneous 5% dextrose injection in patients presenting to the emergency department with low back pain using the visual analog scale (VAS).

The study is planned to include 150 volunteer patients with low back pain who applied to the emergency department of Aksaray University Education and Research Hospital. The patients will be randomly divided into two groups. The first group will receive subcutaneous 5% dextroseprolotherapy (approximately 75 patients), and the second group will receive intramuscular 75 mg diclofenac sodium injection (approximately 75 patients). In all patients, pain intensity will be measured and recorded using the VAS immediately before the injection (baseline), 30 minutes, 1 hour, 2 hours, 12 hours and 24 hours after the injection, and evaluations will be made.

ELIGIBILITY:
* Applying to emergency clinics
* Having isolated low back pain
* Being between the ages of 18-55

Exclusion Criteria:

* Patients under 18 and over 55 years of age,
* intolerance to NSAIDs or allergy to Diclofenac sodium,
* history of gastrointestinal bleeding,
* pregnancy
* patients with red flags for BP (trauma history, recent lumbar surgery, stenosis, spondylolisthesis, lumbar spondylosis with myelopathy)
* documented symptoms as red flags (new leg/foot weakness, new loss of -balance or walking ability, new fever, new night sweats, new urinary retention, new loss of bowel/bladder control)
* known cancer
* long-term steroid use
* patients requiring rescue treatment during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
VAS | In all patients, pain intensity will be measured and recorded using the VAS immediately before the injection (baseline), 30 minutes, 1 hour, 2 hours, 12 hours and 24 hours after the injection, and evaluations will be made.
  It was measured using the Visual Analog Scale (VAS). A score of zero indicated no pain and a score of ten indicated severe, unbearable pain. In all patients, pain intensity will be measured and recorded using the VAS immediately before the injection (baseline), 30 minutes, 1 hour, 2 hours, 12 hours and 24 hours after the injection, and evaluations will be made.

CONTACTS AND LOCATIONS:
Locations (1):
- Aksaray University Education and Research Hospital, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The personal information of the participants in the study will be kept confidential and the data will be shared upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 mount
Access Criteria: Personal information of the participants in the study will be kept confidential and will be provided by the principal investigator if the data is requested for scientific purposes.